CLINICAL TRIAL: NCT06286332
Title: The Effectiveness of Music Therapy on Fatigue and Laboratory Values in Acute Leukemia Patients Undergoing Chemotherapy
Brief Title: Music Therapy in Acute Leukemia Patients With Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University (Other)
Responsible Party: Principal Investigator, Chien-Yu Wu, Nurse, Chang Gung University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Interventional
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Results first posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia; Fatigue
Keywords: AML; Music; Fatigue
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Fatigue | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Therapy (Experimental): Participants received self-selected music app playback for 30 minutes every day and standard therapy. The entire study duration spans 21 days.
  Interventions: Other: Music Therapy
- Standard Care (No Intervention): Participants only received standard care during the entire study duration span of 21 days.

INTERVENTIONS:
Other: Music Therapy — 30 minutes of self-selected music playback every day.
  Arms: Music Therapy

SUMMARY:
The objective of this study is to assess the efficacy of employing music therapy in alleviating fatigue and medical laboratory values among patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
The researchers will explain the study objectives and methods, obtain informed consent, and have participants sign the consent form before commencing the study. Participants are randomly assigned to Group A and Group B. Participants in Group A undergo 30 minutes of self-selected music playback every day in addition to receiving standard therapy, while participants in Group B only receive standard therapy. The entire study duration spans 21 days.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with acute myeloid leukemia by a clinical specialist.
2. Patients undergoing chemotherapy for the first time.
3. Aged 18 years or older, capable of communicating in Mandarin or Taiwanese.
4. Normal hearing ability.
5. No history of psychiatric disorders and clear consciousness.
6. Participants with no prior involvement in any intervention studies related to fatigue management.
7. Demonstrates understanding of the research objectives, willingly participates in the study, and completes the informed consent form.
8. Willing to cooperate with study procedures throughout the research period.

Exclusion Criteria:

1. Severe hearing impairment.
2. Individuals with unstable vital signs or altered consciousness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-01-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Linkou, Taoyuan District, Taiwan, Taiwan

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] AlFayyad I, Al-Tannir M, Yaqub M, Heena H, AlMukaibil N, Ghazwani M, Abu-Shaheen A. Clinically Significant Fatigue in Adult Leukemia Patients: Prevalence, Predictors, and Impact on Quality of Life. Cureus. 2020 Dec 23;12(12):e12245. doi: 10.7759/cureus.12245. PMID 33500864
- [Background] Schumacher A, Wewers D, Heinecke A, Sauerland C, Koch OM, van de Loo J, Buchner T, Berdel WE. Fatigue as an important aspect of quality of life in patients with acute myeloid leukemia. Leuk Res. 2002 Apr;26(4):355-62. doi: 10.1016/s0145-2126(01)00145-x. PMID 11839378
- [Background] Rutkowski S, Czech O, Wrzeciono A, Kiper P, Szczepanska-Gieracha J, Malicka I. Virtual reality as a chemotherapy support in treatment of anxiety and fatigue in patients with cancer: A systematic review and meta-analysis and future research directions. Complement Ther Med. 2021 Sep;61:102767. doi: 10.1016/j.ctim.2021.102767. Epub 2021 Aug 14. PMID 34403772
- [Result] Sezgin MG, Bektas H. The effect of music therapy interventions on fatigue in patients with hematological cancers: a systematic review and meta-analysis of randomized controlled trials. Support Care Cancer. 2022 Nov;30(11):8733-8744. doi: 10.1007/s00520-022-07198-w. Epub 2022 Jun 11. PMID 35689676
- [Result] Burns DS, Azzouz F, Sledge R, Rutledge C, Hincher K, Monahan PO, Cripe LD. Music imagery for adults with acute leukemia in protective environments: a feasibility study. Support Care Cancer. 2008 May;16(5):507-13. doi: 10.1007/s00520-007-0330-z. Epub 2007 Sep 22. PMID 17891547
- [Result] Cassileth BR, Vickers AJ, Magill LA. Music therapy for mood disturbance during hospitalization for autologous stem cell transplantation: a randomized controlled trial. Cancer. 2003 Dec 15;98(12):2723-9. doi: 10.1002/cncr.11842. PMID 14669295
- [Result] Reimnitz L, Silverman MJ. A randomized pilot study of music therapy in the form of patient-preferred live music on fatigue, energy and pain in hospitalized adult oncology patients on a blood and marrow transplant unit. Arts Health. 2020 Jun;12(2):154-168. doi: 10.1080/17533015.2018.1534251. Epub 2018 Oct 18. PMID 31038430
- [Result] Miladinia M, Voss JG, Molavynejad S, Malehi AS, Zarea K, Nouri EM, Ahmadzadeh A. Slow-Stroke Back Massage Compared With Music Therapy for Leukemia-Related Pain and Fatigue: A Randomized Controlled Trial. JCO Oncol Pract. 2021 Nov;17(11):e1614-e1621. doi: 10.1200/OP.21.00156. Epub 2021 Jun 2. PMID 34077243
- [Result] Bates D, Bolwell B, Majhail NS, Rybicki L, Yurch M, Abounader D, Kohuth J, Jarancik S, Koniarczyk H, McLellan L, Dabney J, Lawrence C, Gallagher L, Kalaycio M, Sobecks R, Dean R, Hill B, Pohlman B, Hamilton BK, Gerds AT, Jagadeesh D, Liu HD. Music Therapy for Symptom Management After Autologous Stem Cell Transplantation: Results From a Randomized Study. Biol Blood Marrow Transplant. 2017 Sep;23(9):1567-1572. doi: 10.1016/j.bbmt.2017.05.015. Epub 2017 May 19. PMID 28533058

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with acute myeloid leukemia were recruited from the hematology-oncology ward of a medical center in northern Taiwan.
Groups:
- Experimental: Music Intervention Group: Participants received standard care plus music intervention for 21 days. The music intervention was provided for 30 minutes daily.
- Control: Standard Care Group: Participants received standard care only.
Period: Overall Study
Arm/Group | Experimental: Music Intervention Group | Control: Standard Care Group
Started | 30 | 30
Completed | 27 | 28
Not Completed | 3 | 2
Not completed — Death | 1 | 2
Not completed — Transfer to ICU | 2 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are reported for participants who completed the study and were included in the final analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: Music Intervention Group | Control: Standard Care Group | Total
Number analyzed (Participants) | 27 | 28 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Baseline characteristics are reported for participants who completed the study and were included in the final analysis.
  years | 52.74 (14.04) | 56.43 (14.60) | 54.62 (14.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 24
  Male | 14 | 17 | 31
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Tang Fatigue Rating Scale (Baseline) [Mean (Standard Deviation); unit: scores on a scale] | 135.63 (44.79) | 137.43 (48.23) | 136.55 (46.15)
NRS-11 scores (Baseline) [Mean (Standard Deviation); unit: scores on a scale] — The NRS-11 is a validated, self-reported instrument assessing average fatigue intensity. Scores range from 0 (no fatigue) to 10 (worst possible fatigue). Higher scores indicate a greater level of fatigue.
  scores on a scale | 5.59 (0.36) | 5.40 (0.30) | 5.49 (0.34)
Absolute neutrophil count (ANC) [Mean (Standard Deviation); unit: cells/µL] | 2678.97 (559.50) | 2210.91 (568.45) | 2453.94 (396.29)
Hemoglobin [Mean (Standard Deviation); unit: g/dL] | 8.91 (1.38) | 8.8 (2.03) | 8.86 (1.7)
Albumin [Mean (Standard Deviation); unit: g/dL] | 3.55 (0.47) | 3.51 (0.5) | 3.53 (0.48)

OUTCOME MEASURES:

1. Primary Outcome: Fatigue Score on the Tang Fatigue Rating Scale (TFRS) .
Description: The TFRS is a validated, self-reported instrument assessing average fatigue intensity. It comprises a total of 37 items, with each item rated on a scale of 1 to 10. The total score is calculated by summing all 37 items, resulting in a range of 37 to 370. Higher scores indicate a greater level of fatigue intensity.
Time Frame: Day 21.
Measure: Mean (Standard Deviation); unit: scores
Groups:
- Experimental: Music Intervention Group: Participants received standard care plus music intervention for 21 days.
Arm/Group | Experimental: Music Intervention Group | Control: Standard Care Group
Number analyzed (Participants) | 27 | 28
scores | 106.96 (37.92) | 128.46 (26.32)

2. Secondary Outcome: Absolute Neutrophil Count (ANC) at Day 21.
Description: Absolute neutrophil count (ANC) was assessed through blood samples collected on the 21st day.
Time Frame: Day 21.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | Experimental: Music Intervention Group | Control: Standard Care Group
Number analyzed (Participants) | 27 | 28
cells/µL | 2456.32 (648.11) | 1373.60 (657.88)

3. Secondary Outcome: Hemoglobin Level at Day 21.
Description: Hemoglobin levels were assessed through blood samples collected on the 21st day.
Time Frame: Day 21.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Experimental: Music Intervention Group | Control: Standard Care Group
Number analyzed (Participants) | 27 | 28
g/dL | 9.30 (0.31) | 8.19 (0.16)

4. Secondary Outcome: Albumin Level at Day 21.
Description: Albumin levels were assessed through blood samples collected on the 21st day.
Time Frame: Day 21.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Experimental: Music Intervention Group | Control: Standard Care Group
Number analyzed (Participants) | 27 | 28
g/dL | 3.87 (0.13) | 3.49 (0.14)

5. Primary Outcome: 11-point Numeric Rating Scale (NRS-11).
Description: The NRS-11 is validated, self-reported instrument assessing average fatigue intensity. NRS-11 scores range from 0 (no fatigue) to 10 (worst possible fatigue).
Time Frame: Day 21.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Experimental: Music Intervention Group | Control: Standard Care Group
Number analyzed (Participants) | 27 | 28
scores on a scale | 4.07 (0.38) | 5.00 (0.41)

ADVERSE EVENTS:
Time Frame: From enrollment through study completion (Day 21).
Arm/Group | Experimental: Music Intervention Group | Control: Standard Care Group
All-Cause Mortality (participants affected / at risk) | 1/30 | 2/30
Serious Adverse Events (participants affected / at risk) | 3/30 | 2/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Music Intervention Group (N=30) | Control: Standard Care Group (N=30)
Disease Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Septic shock (Infections and infestations) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-11-14): https://cdn.clinicaltrials.gov/large-docs/32/NCT06286332/Prot_SAP_000.pdf